CLINICAL TRIAL: NCT02097758
Title: Efficacy of Three Dimensional Transesophageal Echocardiography for Percutaneous Device Closure in Atrial Septal Defect
Acronym: ASD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jong-Min Song, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ASD_3D_device size
Record Dates: First submitted 2014-03-25; First posted 2014-03-27 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2023-01

CONDITIONS: Atrial Septal Defect; Successful Device Closure
MeSH Terms: conditions — Heart Septal Defects, Atrial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- transcatheter device closure (Experimental): Choosing device size using three dimensional image and the formula without sizing balloon
  Interventions: Device: Transcatheter device closure

INTERVENTIONS:
Device: Transcatheter device closure — Closure of atrial septal defect with device
  * choosing device size with 3D image and the formula
  * we do not use sizing balloon for choosing of the device size

SUMMARY:
Background: Three-dimensional echocardiographic image for atrial septal defect (ASD) is useful for evaluation of defect size and shape. The investigators suggested optimal device size using three-dimensional transesophageal echocardiographic image and our formula in previous study.

Purpose: In this study, the investigators seek to predict the correct device size and confirm the accuracy of the formula that we made before device closure in ASD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 year-old
* Susceptible indication for atrial septal defect closure
* Potential candidate for device closure

Exclusion Criteria:

* Poor candidate for device closure: multiple ASDs, ect
* Other heart disease requiring open heart surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-03; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Successful device implantation | 1 day

SECONDARY OUTCOMES:
Procedure time | during procedure

OTHER OUTCOMES:
Complications from device | 1 year
  migration or dehiscence of device erosion cardiac rupture

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Min Song, MD PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee PH, Kim GY, Yu JS, Earm I, Kwon KB, Koo HI, Kim TO, Lee S, Sun BJ, Kim DH, Kang DH, Song JK, Song JM. Routine Application of Three-Dimensional Transesophageal Echocardiography-based Device Selection for Transcatheter Closure of Atrial Septal Defect without Balloon Sizing. Eur Heart J Cardiovasc Imaging. 2026 Jan 13:jeag007. doi: 10.1093/ehjci/jeag007. Online ahead of print. PMID 41530892
- [Derived] Jang JY, Heo R, Cho MS, Bae J, Hong JA, Lee S, Ahn JM, Park DW, Kim DH, Kang DH, Song JK, Song JM. Efficacy of 3D transoesophageal echocardiography for transcatheter device closure of atrial septal defect without balloon sizing. Eur Heart J Cardiovasc Imaging. 2018 Jun 1;19(6):684-689. doi: 10.1093/ehjci/jex153. PMID 28633478